CLINICAL TRIAL: NCT05936359
Title: A Phase 1, Open-Label, Multicenter Study of INCA033989 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Myeloproliferative Neoplasms
Brief Title: A Study to Evaluate INCA033989 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCA 33989-101; 2022-502514-86-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-06-21; First posted 2023-07-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Myeloproliferative Neoplasms
Keywords: Myeloproliferative Neoplasms; Ruxolitinib; Myelofibrosis; Essential thrombocythemia; CALR mutation
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1a Dose Escalation Cohort Disease Group A - with MF (Experimental): INCA033989 will be administered at a protocol defined starting regimen in 28-day cycles as monotherapy to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myelofibrosis (MF) will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1a Dose Escalation Cohort Disease Group A - with ET (Experimental): INCA033989 will be administered at a protocol defined starting regimen in 28-day cycles as monotherapy to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with with essential thrombocythemia (ET) will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1a: Dose Escalation Cohort Disease Group B - with TGB-MF SubOpt R (Experimental): INCA033989 will be administered at a protocol defined starting regimen in 28- day cycles and will allow for the evaluation of INCA033989 in combination with ruxolitinib to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myelofibrosis (MF) exhibiting suboptimal response (SubOpt R) will enroll in this group.
  Interventions: Drug: INCA033989; Drug: Ruxolitinib
- Part 1b: Dose Expansion - with MF (Experimental): INCA033989 will be administered as monotherapy at the RDE(s) identified during Part 1a. Participants with treatment group A (TGA) myelofibrosis MF will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1b: Dose Expansion - with TGB-MF SubOpt R (Experimental): INCA033989 will be administered as an add-on therapy in combination with ruxolitinibat at the RDE(s) identified during Part 1a. Participants with treatment Group B (TGB) MF SubOpt R will enroll in this group.
  Interventions: Drug: INCA033989; Drug: Ruxolitinib
- Part 1b: Dose Expansion - with ET (Experimental): INCA033989 will be administered as monotherapy at the RDE(s) identified during Part 1a. Participants with treatment group A (TGA) essential thrombocythemia (ET) will enroll in this group.
  Interventions: Drug: INCA033989
- Part 1c: Dose Expansion (Experimental): INCA033989 will be administered at the dose level found to exhibit an overall positive benefit/risk as monotherapy or as combination therapy with Ruxolitinib. Participants with myelofibrosis (MF) will enroll in this group. The participants enrolled in the monotherapy arm will be offered the option to crossover to combination therapy with ruxolitinib if a suboptimal response to monotherapy is observed after 12 weeks.
  Interventions: Drug: INCA033989; Drug: Ruxolitinib

INTERVENTIONS:
Drug: INCA033989 — INCA033989 will be administered at protocol defined dose.
Drug: Ruxolitinib — Rux will be administered according to Prescribing Information/SmPC.
  Other Names: Jakafi
  Arms: Part 1a: Dose Escalation Cohort Disease Group B - with TGB-MF SubOpt R; Part 1b: Dose Expansion - with TGB-MF SubOpt R; Part 1c: Dose Expansion

SUMMARY:
This study is being conducted to evaluate the safety, tolerability, and dose-limiting toxicity (DLT) and determine the maximum tolerated dose (MTD) and/or recommended dose(s) for expansion (RDE) of INCA033989 administered as a monotherapy or in combination with ruxolitinib in participants with myeloproliferative neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 6 months.
* Willingness to undergo a pretreatment and regular on-study BM biopsies and aspirates (as appropriate to disease).
* Existing documentation from a qualified local laboratory of CALR exon-9 mutation.
* Participants with MF and ET as defined in the protocol.

Exclusion Criteria:

* Presence of any hematological malignancy other than ET, PMF, or post-ET MF.
* Active invasive malignancy over the previous 2 years.
* Active HBV/HCV, HIV.
* History of clinically significant or uncontrolled cardiac disease.
* Has undergone any prior allogenic or autologous stem-cell transplantation or such transplantation is planned.
* Laboratory values outside the Protocol-defined ranges.
* Participants undergoing treatment with G-CSF, GM-CSF, or TPO-R agonists at any time within 4 weeks before the first dose of study treatment.
* Prior history of major bleeding, or thrombosis within the last 3 months prior to study enrollment.
* Any prior chemotherapy, immunomodulatory drug therapy, immunosuppressive therapy, biological therapy, endocrine therapy, targeted therapy, antibody, or hypomethylating agent used to treat the participant's disease within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* For TGBs only: Undergoing treatment with a potent/strong inhibitor or inducer of CYP 3A4/5 within 14 days or 5 half-lives (whichever is longer) before the first dose of study treatment, or expected to receive such treatment during the study.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 3 years and 60 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug monotherapy and in combination with ruxolitinib
Number of participants with TEAEs leading to dose modification or discontinuation | Up to 3 years and 60 days
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
Participants with MF: Response using the revised IWG-MRT and ELN response criteria for MF | Up to 3 years and 60 days
  Defined as the percentage of participants with Response using the revised IWG-MRT and ELN response criteria.
Participants With MF: Percentage of participants achieving spleen volume reduction as defined in the protocol | Up to 3 years and 60 days
  Defined as percentage of participants with a protocol defined Spleen Volume Reduction.
Participants with MF with symptomatic anemia: Anemia Response | Up to 3 years and 60 days
  For non transfusion-dependent (TD) participants: An Hb increase relative to baseline as defined in the protocol if non-TD at baseline. For TD participants: Achieving transfusion independency (TI) as defined in the protocol.
Participants With ET: Response Rate | Up to 3 years and 60 days
  Defined as the proportion of participants with Complete Response or Partial Response when treated with study drug.
Participants With ET: Mean change from baseline of total symptom score (TSS) | Up to 3 years and 60 days
  Mean change of TSS from baseline.
Mean change in disease-related allele burden | Up to 3 years and 60 days
  Mean change in disease-related allele burden.
Pharmacokinetics Parameter: Cmax of INCA33989 | Up to 3 years and 60 days
  Defined as maximum observed plasma concentration of INCA33989.
Pharmacokinetics Parameter: Tmax of INCA033989 | Up to 3 years and 60 days
  Defined as the time to reach the maximum plasma concentration of INCA33989.
Pharmacokinetics Parameter: Cmin of INCA33989 | Up to 3 years and 60 days
  Defined as the minimum observed plasma concentration of INCA33989.
Pharmacokinetics Parameter: AUC(0-t) of INCA33989 | Up to 3 years and 60 days
  Defined as the area under the concentration-time curve up to the last measurable concentration of INCA33989.
Pharmacokinetics Parameter: AUC 0-∞ of INCA33989 | Up to 3 years and 60 days
  Defined as the area under the concentration-time curve from 0 to infinity of INCA33989.
Pharmacokinetics Parameter: CL/F of INCA33989 | Up to 3 years and 60 days
  Defined as the apparent oral dose clearance of INCA33989.
Pharmacokinetics Parameter: Vz/F of INCA33989 | Up to 3 years and 60 days
  Defined as the apparent oral dose volume of distribution of INCA33989.
Pharmacokinetics Parameter: t1/2 of INCA33989 | Up to 3 years and 60 days
  Defined as the apparent terminal phase disposition half-life of INCA33989.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (29):
- Australia (4):
  - Royal Brisbane and Women'S Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Qc, Montreal, Quebec
- Denmark (3):
  - Odense University Hospital, Odense C
  - Sjaellands Universitetshospital, Roskilde
  - Vejle Hospital, Vejle
- France (4):
  - Institut Bergonie, Bordeaux
  - Chu Nimes, Nîmes
  - Hospital Saint Louis, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - University Medical Center Rwth Aachen, Aachen
  - Universitatsklinikum Halle (Saale), Halle
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - Aou Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
- Japan (5):
  - National Cancer Center Hospital East, Chiba-ken
  - Kagoshima University Hospital, Kagoshima
  - Osaka Metropolitan University Hospital, Osaka
  - Nippon Medical School Hospital, Tokyo
  - Mie University Hospital, Tsu
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari I Politecnic La Fe, Valencia
- United Kingdom (3):
  - Guys and St Thomas Nhs Foundation Trust, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate INCA033989 Administered as a Monotherapy or in Combination With Ruxolitinib in Participants With Myeloproliferative Neoplasms — https://www.incyteclinicaltrials.com/study/?id=INCA%2033989-101&SearchTerm=INCA%2033989-101&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=